CLINICAL TRIAL: NCT00583297
Title: Identifying Genetic Markers That Predict Microvolt T-wave Alternans Status and Arrhythmia Risk in Patients With Ischemic Heart Disease
Brief Title: Genetic Substudy of the Alternans Before Cardioverter Defibrillator (ABCD) Trial
Acronym: ABCD
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000001; ABCD (Other: CardioDx)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2017-10

CONDITIONS: Ventricular Tachycardia; Cardiovascular Diseases; Arrythmia; CVD
Keywords: Arrhythmia; Heart Failure; T-wave Alternans; Implanted Cardioverter Defibrillator; Biological Markers; Molecular Genetics; Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CVD; Precision Medicine; Sudden Cardiac Death; Electrophysiology Study; Cardiovascular Disease; ICD; EPS; SCD; TWA
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiovascular Diseases; Arrhythmias, Cardiac; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and saliva.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ABCD Subjects: The cohort will consist of original subjects of the ABCD trial who consent to participate in the genetic sub-study

SUMMARY:
The ABCD clinical study (ClinicalTrials.gov Identifier NCT00187291) was designed to determine if a T-Wave Alternans (TWA) test is equivalent to an Electrophysiology Study (EPS) in predicting life-threatening heart rhythms in patients with ischemic heart disease, left ventricular dysfunction, and non-sustained tachycardia. The purpose of the ABCD Genetic sub-study is to identify genetic markers that predict TWA status and arrhythmia risk in this same population.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that therapy directed primarily by a T wave alternans (TWA) test, measured non-invasively during exercise, is equivalent to therapy directed by an electrophysiological study (EPS) in predicting spontaneous ventricular tachyarrhythmic events (VTEs) in patients with ischemic heart disease, left ventricular dysfunction, and asymptomatic non-sustained ventricular tachycardia (NSVT). In the absence of any previous life-threatening ventricular arrhythmia (i.e., for primary prevention), ICD implantation is currently indicated in patients with ischemic heart disease, left ventricular dysfunction, asymptomatic non-sustained ventricular tachycardia, and a positive EPS. The objective of this study is to demonstrate that a TWA test directed therapy is equivalent to EPS directed therapy in guiding ICD implantation for the purpose of primary prevention of sudden cardiac death (SCD) in patients with ischemic heart disease, left ventricular dysfunction, and asymptomatic non-sustained ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

Subjects previously enrolled in the ABCD trial sponsored by St. Jude Medical (ClinicalTrials.gov Identifier NCT00187291)

* patients with ischemic heart disease
* left ventricular ejection fraction (LVEF) < 40%
* non-sustained ventricular tachycardia

Exclusion Criteria:

Individuals who were not previously enrolled in the ABCD trial are not eligible for this genetic sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the ABCD genetic sub-study includes all living individuals currently enrolled in the ABCD trial (total study enrollment=629; 566 analyzed in the trial) Participants of the ABCD trial underwent TWA and EPS testing to determine their risk for ventricular arrhythmia and most have received an implantable cardioverter defibrillator (ICD). The ABCD trial collected extensive longitudinal clinical data including medical and medication histories, incidence of ventricular arrhythmias, defibrillator shocks, other cardiovascular events, and mortality.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Genotype and Pre-implant T-wave alternans status. | two years as per original ABCD trial
  Genotype and Pre-implant T-wave alternans status.

SECONDARY OUTCOMES:
Genotype and occurrence of appropriate cardioversion | two years per original ABCD trial
  Genotype and occurrence of appropriate cardioversion for ventricular tachycardia or ventricular fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Sehnert, MD, Study Director — CardioDx, Inc.; Elizabeth Kaufman, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Wilson LD, Wan X, Rosenbaum DS. Cellular alternans: a mechanism linking calcium cycling proteins to cardiac arrhythmogenesis. Ann N Y Acad Sci. 2006 Oct;1080:216-34. doi: 10.1196/annals.1380.018. PMID 17132786
- [Background] Bloomfield DM, Bigger JT, Steinman RC, Namerow PB, Parides MK, Curtis AB, Kaufman ES, Davidenko JM, Shinn TS, Fontaine JM. Microvolt T-wave alternans and the risk of death or sustained ventricular arrhythmias in patients with left ventricular dysfunction. J Am Coll Cardiol. 2006 Jan 17;47(2):456-63. doi: 10.1016/j.jacc.2005.11.026. Epub 2005 Dec 15. PMID 16412877